CLINICAL TRIAL: NCT04170816
Title: Comparing Dry Needling With And Without Kinesio Taping® in The Treatment of Non-Specific Chronic Low Back Pain
Brief Title: Dry Needling With And Without Kinesio Taping® in The Non-Specific Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kars State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Bagcier, Principal Investigator, Kars State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80576354-050-99/167
Record Dates: First submitted 2019-09-15; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Non-Spesific Chronic Low Back Pain
Keywords: Dry needling; Kinesiotape; Low-back pain
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling; Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DN plus KT group (Active Comparator): DN plus KT therapy is going to be applied 3 sessions in 1-week intervals. Dry Needling Theraphy: DN therapy is going to be applied on active myofascial trigger points (MTrP) in quadratus lumborum, gluteus medius and lumbar multifidus muscles.
  Kinesio Taping Application: Tapes is going to be left on the patient's body for 5 days.
  Interventions: Device: Dry needling
- DN group (Active Comparator): DN will be applied 3 sessions in 1-week intervals. Dry Needling Theraphy: DN therapy was applied on active myofascial trigger points (MTrP) in quadratus lumborum, gluteus medius and lumbar multifidus muscles.
  Interventions: Device: Dry needling

INTERVENTIONS:
Device: Dry needling — DN and KT therapy will be applied 3 sessions in 1-week intervals
  Other Names: Kinesiotape

SUMMARY:
We wiil evaluate the efficiency of adding kinesio taping (KT) therapy to dry needling (DN) therapy on pain, functionality and depression parameters in 60 patients with nonspecific chronic low back pain (nCLBP).

DETAILED DESCRIPTION:
A total of 60 patients will be included in the study. 30 patients will be in the treatment group and 30 patients will be in the control group. Both groups will be underwent 3 sessions with 1-week intervals on active myofascial trigger points in lumbar multifidus, quadratus lumborum and gluteus medius muscles in DN therapy. KT application will be performed after every DN session in the study group. Pain will evaluate with visual analog scale, functionality was evaluated with Oswestry Disability Index and the status of depression will be evaluated with Beck Depression Index before the treatment and at the first month.

ELIGIBILITY:
Inclusion Criteria:

* having no abnormal results in routine blood tests
* having no known acute or chronic inflammatory disease
* an education level required for understanding the applied treatment, interventions

Exclusion Criteria:

* malignancies
* active infection
* history of common inflammatory rheumatic disease
* trauma in spinal area, skin lesion, presence of infection or open wounds
* radiculopathy
* peripheral circulation disorder
* use of warfarin due to coagulopathy
* arthropathy
* congenital or acquired spinal pathology
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold | 3 week
  Amount of pressure (Kg/cm2) applied at the lomber multifidus muscle, quadratus lumborum and gluteus medius muscle myofascial trigger point site that elicit pain for the patient will be reported
Pain by visual analog scale (VAS) | 3 week
  Visual analog scale (VAS,0-10) will be used to assess resting, activity and night pain.
Oswestry disability Index (ODI) | 3 week
  Changes from the Baseline, ODI is an effective tool to provide information on the extent of backache affecting the patient ability to cope with tasks of everyday life. Ten sections are included in the ODI tool with a total possible score of 5 for each section. The first statement carries a score of 0, and the last has a score of 5.
Beck Depression Inventory | 3 week
  This is a 21-item standard assessment used to measure clinical depression. Scores on this assessment range from 0 to 63, where higher scores indicate higher levels of depression.